CLINICAL TRIAL: NCT06932575
Title: The Effect of Andullation Therapy on Pain and Anxiety After Oocyte Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Tuğba Kartal, Assistant Professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-80558721-050.99-154981
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Pain Management; Anxiety Management; Oocyte Retrieval
Keywords: Infertility; Oocyte Retrieval; Andullation; Pain; Anxiety
MeSH Terms: conditions — Agnosia; Infertility; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group received andullation therapy (Experimental): The experimental group received andullation therapy for 30 minutes using an andullation therapy bed after oocyte retrieval
  Interventions: Device: Andullation Therapy Bed
- The control group only applied scales (No Intervention): The control group did not receive andullation therapy after oocyte retrieval.

INTERVENTIONS:
Device: Andullation Therapy Bed — andullation therapy applied for 30 minutes after oocyte retrieval
  Arms: The experimental group received andullation therapy

SUMMARY:
The goal of this clinical trial is to evaluate the effect of andullation therapy in the management of pain and anxiety that occur in the patient follow-up after oocyte retrieval. The main questions it aims to answer are:

* Does andullation therapy after oocyte retrieval reduce pain measured immediately after the end of therapy?
* Does andullation therapy after oocyte retrieval reduce anxiety measured immediately after the end of therapy?

Researchers will compare experimental and control groups to see if andullation therapy reduce pain and anxiety after oocyte retrieval.

Participants will:

* Take State Anxiety Inventory before oocyte retrieval.
* Take andullation therapy or not after oocyte retrieval
* Take the State Anxiety Inventory and Visual Analog Scale at 1 hour, 1.5 hours, 6 hours, and 24 hours after oocyte retrieval.

DETAILED DESCRIPTION:
During the oocyte retrieval procedure, midazolam, propofol, and remifentanil were administered intravenously by the anesthesia technician at doses determined by the anesthesiologist. During the two-hour period in which the women were closely monitored the procedure, 1 g of paracetamol vial recommended by the physician was administered intravenously by a reproductive health nurse to the women who stated that they had a lot of pain. Medical and technical details about the procedure and the patient, including the sedation protocol applied during oocyte retrieval, the number of oocytes collected, and whether a painkiller was administered was determined by the researcher based on information obtained from the physician and the patient's medical records.

In this study, the P05 relaxation program, one of the 10 different health programs of the andullation therapy bed, was used. Using the device control, the regional vibration intensity was set to 4, ensuring consistency across all regions. Infrared heat was activated in the neck and spine area with the H1 button and in the leg area with the H2 button. With this program, it was aimed to reduce anxiety by providing deep relaxation in the body and to provide the necessary energy for the body to repair itself.

to clearly show the duration of the effect of andullation therapy on pain and anxiety, intermittent scale applications were performed starting from before oocyte retrieval, when anxiety was thought to be the highest, until 24 hours after oocyte retrieval, when we expected the pain to gradually disappear.

ELIGIBILITY:
Inclusion Criteria:

* Having an oocyte retrieval procedure regardless of the cause of infertility,
* Being at least literate,
* Being between the ages of 18-49,
* Accepting to participate in the study,
* Pain level above 0, as measured by the VAS scale, applied after the oocyte retrieval procedure.

Exclusion Criteria:

* Having chronic pain problems,
* Having communication problems,
* Having any nervous or musculoskeletal disorders that would prevent them from lying flat on the massage bed,
* Having any diagnosed psychiatric illness,
* Refusal to participate in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Pain Severity after Oocyte Retrieval | 1, 1.5, 6, and 24 hours after oocyte retrieval
  Measure the relationship between pain severity in experimental and control groups after oocyte retrieval using Visual Analog Scale. In a 10-point VAS scoring: 0 indicates no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain, and 7-10 indicates severe pain

SECONDARY OUTCOMES:
Anxiety Level after Oocyte Retrieval | 1, 1.5, 6, and 24 hours after oocyte retrieval
  Measure the relationship between anxiety level in experimental and control groups after oocyte retrieval using State Anxiety Inventory. The lowest score to be obtained from the scale is 20, and the highest score is 80. A cut-off score of 40 is commonly used to define possible levels of clinical anxiety. The higher the score on the scale, the higher the level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. VEHBİ YAVUZ TOKGÖZ, Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Eskişehir, Turkey (Türkiye)